CLINICAL TRIAL: NCT00236405
Title: A Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Effects of of PROCRIT� (Epoetin Alfa) on Short-Term Outcomes in Orthopedic Subjects Undergoing Primary Unilateral Knee Arthroplasty
Brief Title: PROCRIT and Short-Term Outcomes in Orthopedic Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to poor enrollment.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003193
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Surgery, Arthroscopy
Keywords: Anemia; erythropoetin; quality-of-life outcomes
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to compare the effect of perioperative administration of PROCRIT to that of autologous blood donation on post-operative rehabilitation outcomes in patients undergoing unilateral knee surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effect of perioperative administration of PROCRIT to that of preoperative autologous donation on post-operative rehabilitation outcomes in subjects undergoing primary unilateral knee arthroplasty.

Secondary objectives are : 1) To compare the effect of perioperative administration of PROCRIT to that of preoperative autologous donation on hemoglobin, change in hemoglobin, number of units transfused and transfusion rate during the study period; and 2) To compare the effect of perioperative administration of PROCRIT to that of preoperative autologous donation on inpatient rehabilitation length of stay.

The study will test the hypothesis that perioperative administration of PROCRIT will improve post-operative rehabilitation outcomes, compared with preoperative autologous donation. 40,000U PROCRIT or Placebo SC in relation to surgery date: Days -21, -14, -7, 0 (day of surgery), 7, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for primary unilateral knee arthroplasty with an expected discharge into an inpatient rehabilitation facility
* Hemoglobin >11 to <13 g/dL at screening and preoperative day -21
* Age 18 years or older
* Female subjects must be post-menopausal for at least one year or surgically sterile (hysterectomy or tubal ligation). Women of childbearing age must have negative pregnancy test(s) (serum HCG RIA at screening and urine at preoperative day -21, if applicable
* Preoperative lead time of at least 21 days

Exclusion Criteria:

* Medical conditions including: Known iron deficiency (defined as serum ferritin <50 mg/l)
* chronic renal failure, significant hematological disease, uncontrolled hypertension, new onset seizures/uncontrolled seizures
* Expected to need another lower extremity major joint replacement within six months
* Undergoing cancer chemotherapy
* History of thrombotic vascular events including but not limited to stroke, transient ischemic attack, myocardial infarction and deep venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-03; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in composite FIM scores (from entry into the inpatient rehabilitation facility to discharge from inpatient rehabilitation) divided by the LOS, denoted as DFIM/LOS, or "rate of functional recovery".

SECONDARY OUTCOMES:
LOS in the inpatient rehabilitation facility; Total FIM score; FIM Physical Sub-score LASA score; FACIT-An score. Safety evaluations include the incidence of adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Procrit (Epoetin alfa) on Short-Term Outcomes in Orthopedic Subjects Undergoing Primary Unilateral Knee Arthroplasty — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=505&filename=CR003193_CSR.pdf